CLINICAL TRIAL: NCT05219760
Title: LIVIA 2.0: A Randomized Controlled Trial of Two French Internet Intervention for Adults Struggling With Prolonged Grief Symptoms After the Loss of a Close One (by Bereavement or Separation/Divorce)
Brief Title: LIVIA 2.0 : A RCT Of Two French Internet Intervention For Adults Struggling With Prolonged Grief Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Debrot Anik (Other)
Responsible Party: Sponsor-Investigator, Debrot Anik, Sponsor-Investigator, University of Lausanne
Organization: University of Lausanne (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-D0086
Record Dates: First submitted 2021-12-23; First posted 2022-02-02 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Prolonged Grief Disorder
MeSH Terms: conditions — Prolonged Grief Disorder

STUDY DESIGN:
Intervention Model Description: The study aim to compare the efficacy of an IBI targeting complicated grief symptoms (LIVIA 2.0) compared to an already investigated IBI (LIVIA 1) using a guidance on demand design in a randomised controlled trial.
  Both programs are composed of 10 weekly sessions proposing educational material, questionnaires and exercises. They are based on current scientific theories of grief but present their content differently. Compared to LIVIA 1, LIVIA 2.0 is less based on academic readings and participants can choose more freely which topics and exercises they want to do. LIVIA 2.0 also offers a system of reminder messages to maximize adherence as well as more elaborate automated guidance.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LIVIA 1 (Active Comparator): LIVIA 1 is a 12-week intervention composed of 10 sessions, whereby we recommend completing one session per week. It includes psychoeducational content and exercises that are based on empirically validated intervention tools, mainly issued from Cognitive-Behavioral Therapy.
  Interventions: Device: LIVIA
- LIVIA 2.0 (Experimental): LIVIA 2.0 is a 12-week intervention composed of 10 sessions, whereby we recommend completing one session per week. It includes psychoeducational content and exercises that are based on empirically validated intervention tools, mainly issued from Cognitive-Behavioral Therapy but also from positive psychology and cognitive psychopathology frame.
  Interventions: Device: LIVIA

INTERVENTIONS:
Device: LIVIA — The study aim to compare the efficacy of an IBI targeting complicated grief symptoms (LIVIA 2.0) compared to an already investigated IBI (LIVIA 1) using a guidance on demand design in a randomised controlled trial.
  Both programs are composed of 10 weekly sessions proposing educational material, questionnaires and exercises. They are based on current scientific theories of grief but present their content differently. Compared to LIVIA 1, LIVIA 2.0 is less based on academic readings and participants can choose more freely which topics and exercises they want to do. LIVIA 2.0 also offers a system of reminder messages to maximize adherence as well as more elaborate automated guidance.

SUMMARY:
The investigators aim to compare the efficacy of an IBI targeting complicated grief symptoms (LIVIA 2.0) compared to an already investigated IBI (LIVIA 1) using a guidance on demand design in a randomised controlled trial (RCT).

More specifically, the investigators will test the following primary hypotheses:

* Both interventions will significantly increase participants' well-being and decrease their distress, and those changes will be stable until follow-up.
* LIVIA 2.0 will be more efficient than LIVIA 1 on all measure outcomes.
* LIVIA 2.0 will have less dropouts than LIVIA 1.

DETAILED DESCRIPTION:
Secondary objectives are the following:

* Participants of LIVIA 2.0 will require less guidance (number of people requesting support and number of e-mails exchanged) than participants in LIVIA 1. The investigators will also explore which session triggers more requests of guidance.
* Using a monitoring of participants' state throughout the completion of the programme in LIVIA 2.0, the investigators will explore the short-term efficacy of each module on participants' weekly mood, solitude feelings and grief symptoms.
* The investigators will compare participants' satisfaction in both versions of LIVIA.
* The investigators will also explore the role of attachment style, type of loss, relationship quality with the partner, the interpersonal closeness with the lost person, symptom severity and level of solitude at onset as moderators of the efficacy of the programmes.
* The investigators will explore the semantic content of the exercises included in the programme to see if this is related with the improvement over the assessment period.

ELIGIBILITY:
Inclusion Criteria:

* Bereavement or separation/divorce
* Either of these events should have happened more than 6 months before participating in the study
* Feeling the need for support to cope with the loss (a diagnosis of complicated grief is not necessary)
* Age: 18 years or older
* Regular Internet access
* Mastery of the French language - Approved ICF

Exclusion Criteria:

* Moderate to acute current suicidality (SIDAS > 19)
* Severe psychological or somatic disorders which need immediate treatment.
* Concomitant psychotherapy
* Prescription or change in dosage of psychoactive drugs in the month prior or during the self-help intervention.
* Inability to follow the procedures of the study, e.g. due to comprehension problems
* Enrolment of the investigator, his/her family members, employees, and other dependent persons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-05-06 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Change in complicated grief symptoms | Pretest; 12-week post-test; 3-month Follow-up
  assessed with a French version (Cherblanc & Zech, 2021) of The Traumatic Grief Inventory (Boelen et al., 2019), on a scale ranging from 1 = never to 5 = always. The mean score is used as a final score. Higher score represent a higher symptom load.
Change in depression symptoms | Pretest; 12-week post-test; 3-month Follow-up
  assessed with the Patient Health Questionnaire-9 (Kroenke & Spitzer, 2002; Kroenke, Spitzer & Williams, 2001), on a scale ranging from 0 = never to 4 = practically every day. The sum of the scores is used as a final score. Higher score represent a higher symptom load.
Change in well-being | Pretest; 12-week post-test; 3-month Follow-up
  measured with the French version (Villieux et al., 2016) of the Flourishing Scale (Diener et al., 2010), on a scale ranging from 1 = I completely disagree, to 7 = I completely agree. The mean score is used as a final score. Higher score represent a better psychological well-being.

SECONDARY OUTCOMES:
Change in anxiety symptoms | Pretest; 12-week post-test; 3-month Follow-up
  assessed with the Generalized Anxiety Scale (Micoulaud-Franchi et al., 2016; Spitzer et al., 2006), on a scale ranging from 0 = never to 4 = practically every day. The sum of the scores is used as a final score. Higher score represent a higher symptom load.
Change in grief coping strategies | Pretest; 12-week post-test; 3-month Follow-up
  measured with the Coping with Bereavement Questionnaire (Ryckebosch-Dayez et al., 2016), on a scale ranging from 1 = almost never to 5 = always. Higher scores represent a higher use of the coping strategy.
Change in aspects related to identity | Pretest; 12-week post-test; 3-month Follow-up
  Measured with three scales:
  1. The Self-Concept Clarity (Brunot et al., 2015; Campbell et al., 1996) has a scale ranging from 1 = I completely disagree to 5 = I completely agree. The mean score is used as a final score. Higher score represent a lesser clarity of the self-concept.
  2. The Centrality of Event Scale (Berntsen & Rubin, 2006; Ceschi et al., 2009) has a scale ranging from 1 = I completely disagree to 5 = I completely agree. The mean score is used as a final score. Higher score represent a higher centrality of the event of loss.
  3. Questions about self-continuity (Lampraki et al., 2019), on a scale ranging from 1 = does not suit me to 5 = suits me perfectly. The mean score is used as a final score. Higher score represent a higher self-continuity.
Satisfaction with the program (utility, clarity, impact, etc.) assessed by an adapted version of the CSQ-I | 12-week post-test
  The investigators will measure the satisfaction with the program, by using a translated and adapted version of the Client Satisfaction Questionnaire (CSQ-I; Boß et al., 2016) assessing different quantitative and qualitative questions. These questions will be evaluated separately.
Change in the monitoring of the mood, solitude feelings and grief symptoms | Days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, 85
  The investigators will weekly monitor the mood of the participants of LIVIA 2 using a single item ("How would you describe your current mood" on a scale ranging from 0 (very bad) to 6 (very good). Moreover, the investigators will weekly monitor the grief and solitude symptoms on a scale ranging from 1 (strongly disagree) to 5 (strongly agree) with the following items: "During the past 24 hours: (1) I have felt negative emotions ; (2) I have had negative images or thoughts ; (3) I felt blocked in my behaviour (what I do, my activities) ; (4) I felt lonely ; (5) I felt like I had a clear sense of who I am and what I want in life.
Indicators of verbal immediacy (use of first-person pronouns and present tense words) and so-called "we-talk" (first-person plural pronouns) | 12-week Post-test
  The investigators will analyse the linguistic behaviours and the semantic content in the exercises where the participants are required to describe a situation related to the loss. The objective is to test if some semantic categories (e.g. "we-talk", Bourassa et al., 2018) are associated with the efficacy of the programme.
Degree of required guidance in each group | 12-week Post-test
  number of participants requiring guidance and number of e-mails exchanged

CONTACTS AND LOCATIONS:
Overall Officials: Valentino Pomini, Principal Investigator — University of Lausanne
Locations (1):
- University of Lausanne - Institute of Psychology, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
After publishing the results, the investigators will make the codified data available on request.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Access Criteria: The investigators demand that the purpose of the request is clearly stated.

REFERENCES:
- [Derived] Debrot A, Efinger L, Kheyar M, Pomini V, Berthoud L. A French-Language Web-Based Intervention Targeting Prolonged Grief Symptoms in People Who Are Bereaved and Separated: Randomized Controlled Trial. JMIR Form Res. 2024 Oct 16;8:e57294. doi: 10.2196/57294. PMID 39412869
- [Derived] Debrot A, Kheyar M, Efinger L, Berthoud L, Pomini V. Supporting People Who Have Lost a Close Person by Bereavement or Separation: Protocol of a Randomized Controlled Trial Comparing Two French-Language Internet-Based Interventions. JMIR Res Protoc. 2022 Jun 23;11(6):e39026. doi: 10.2196/39026. PMID 35737454
- See also: Website of the program — https://psyconsultonline.ch/